CLINICAL TRIAL: NCT06469515
Title: Enhanced Continuity of Postoperative Care for Older People in Their Neurocognitive Recovery After Cardiac Surgery
Brief Title: Older People's Neurocognitive Recovery After Cardiac Surgery
Acronym: ECPON
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lina Bergman, Principal Investigator, Karolinska Institutet
Other Study IDs: 2023-02089
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Recovery; Cardiac Surgery
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Elective or urgent cardiac surgery — This is a longitudinal observational study to explore postoperative cognitive recovery among older persons (aged 65 or older) undergoing elective or urgent cardiac surgery via sternotomy.

SUMMARY:
Society is aging and advantages in anesthesia and surgery allow more complex interventions in older persons. Old age is a significant risk factor for the development of postoperative neurocognitive decline characterized by a gradual decrease in performance in several cognitive domains such as memory, attention, information processing, and executive functions, leading to problems with performing daily activities and maintaining independence and postoperative complications. The purpose of this study is to measure older persons' postoperative neurocognitive function, to detect neurocognitive decline, and to identify risk factors and difficulties in daily living as well as explore close relatives' experiences of it. We will include 220 participants ≥65 years of age undergoing planned cardiac surgery. Cognitive symptoms and signs and neurocognitive function will be assessed up to 6 months after surgery. Risk/affected factors such as delirium, functional status, recovery, depression, and healthcare-related quality of life, as well as close relative's experiences and burden, will be measured. The results will have immediate relevance for a substantial number of older persons undergoing surgery, and their close relatives, by enhancing knowledge about postoperative cognitive decline and recovery, and subsequently identifying what support needs to be implemented.

DETAILED DESCRIPTION:
The overarching purpose of the study is to investigate cognitive function, symptoms, and complaints after cardiac surgery among individuals aged 65 and older, as well as to describe the experiences and perspectives of close relatives regarding the same phenomena. The study is expected to answer the following scientific research questions:

1. What is the incidence of postoperative cognitive decline and the occurrence of cognitive symptoms and complaints in older individuals up to 6 months after cardiac surgery?
2. Is there a correlation between preoperative cognitive status and postoperative cognitive decline, and if so, which cognitive function (executive function, attention, memory) is most affected?
3. Is there any correlation between postoperative delirium and postoperative cognitive decline, and if so, which cognitive function is most affected?
4. Which factors (such as age, operation time, perceived self-efficacy, frailty, and depression) affect the risk of suffering from postoperative cognitive decline?
5. Is postoperative cognitive decline associated with increased symptom burden, impaired functional level, fatigue, frailty, deteriorated quality of life, and an increased number of unplanned contacts with healthcare services?
6. How do older individuals experiencing cognitive symptoms and complaints perceive their postoperative recovery and return to daily life?
7. How do close relatives perceive the patient's postoperative cognitive function, recovery, and return to everyday life, and how does this affect the relative's own life?

The study is a longitudinal observational study with a mixed-method approach planned to be conducted at two thoracic surgical units in Sweden. In total, 220 patients and one of their relatives are planned to be included and followed up for 6 months after undergoing cardiac surgery. The study will be reported following the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) guidelines.

In connection with the decision on surgery, it is assessed whether the patient is suitable for inclusion. Potential study participants will receive written and verbal information about the study and will then be asked to participate. After the participant has given informed written consent, baseline data will be collected. This can be done digitally, through home visits, or at the hospital. Included patients will be asked if they have any relatives who can be approached for participation. Potential study participants (relatives) will then be informed about the study and subsequently asked for participation. Baseline data from relatives is collected before the time of surgery.

Enrolled participants (patients) will undergo neurocognitive testing before and at 1, 3, and 6 months after surgery. Mindmore-P is a digitized test battery designed to measure cognitive function. The battery consists of four tests that assess various cognitive functions, including verbal episodic memory, executive function, attention, and processing speed. Mindmore-P is tailored for independent administration via a computer. The tests are conducted through a digital platform (CE-certified) that also contains normative data. All other questionnaires can be answered either electronically or in paper format. During their hospital stay, included participants will be assessed for postoperative delirium.

Descriptive data are presented with mean, median, frequency/proportion, and appropriate measures of dispersion. Postoperative cognitive dysfunction is defined as the patient deviating one standard deviation from the baseline measurement on at least two of the cognitive tests included in the cognitive test battery. Individual data are adjusted against a norm database to control for variation and learning effects. Comparisons between groups will be made using parametric and non-parametric tests based on data level and normal distribution. Associations and relationships will be examined with logical multivariate regression models. Qualitative data will be analyzed with content analysis. Mixed-method analysis may be appropriate to triangulate and compare qualitative and quantitative data to best answer certain scientific questions.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective or urgent open-heart surgery or minimally invasive cardiac surgery
* Resident in the area/region for the current thoracic clinic
* Able to read and understand Swedish

Exclusion Criteria:

* Physical, mental, and cognitive difficulties that prevent the individual from completing the cognitive tests
* Undergone surgery within the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of patients (65 years or older) who have undergone cardiac surgery and their relatives. The study participant is qualified for inclusion if he or she meets all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive complaints | Before surgery and weekly up to three months after surgery
  The Swedish Quality of Recovery cognitive version (SwQoR-Cog) is a self-assessment questionnaire that measures postoperative symptoms. The form consists of 14 statements regarding symptoms and discomforts, of which 11 address cognitive symptoms and 3 are related to pain and nausea. Symptoms and discomforts are rated on an 11-point scale (0=not at all to 10=all the time).
Changes in postoperative cognitive function, part 1 | Before surgery and 1, 3, and 6 months after surgery
  Consortium to Establish a Registry for Alzheimer´s Disease (CERAD) A 10-word verbal learning test with 3 learning trials, a recall trial after ~7 min.
Changes in postoperative cognitive function, part 2 | Before surgery and 1, 3, and 6 months after surgery
  Trail Making Test (TMT- A & B) consists of 25 circles with letters or numbers on the screen.
Changes in postoperative cognitive function, part 3 | Before surgery and 1, 3, and 6 months after surgery
  Stroop Colour-Word Test (SCW). 24 words spelling out the name of a colour which is printed in contrasting ink colours (e.g., the word "green" printed with red ink), and the participant is asked to tell the printed colour of the word rather than the word rather than the actual meaning of the word.
Changes in postoperative cognitive function, part 4 | Before surgery and 1, 3, and 6 months after surgery
  Symbol Digits Processing Test (SDPT). The test consists of nine symbol-digit pairings at the top of the screen, one symbol in the middle of the screen, and a number grid at the bottom.

SECONDARY OUTCOMES:
Postoperative delirium | Twice daily up to postoperative day 7
  The Nursing Delirium Scale (Nu-DESC) is an assessment scale where five symptoms are identified and evaluated. A total score of ≥ 2 points indicates the presence of delirium.
Perceived self-efficacy | Before surgery and 1, 3, and 6 months after surgery
  The Swedish General Self-Efficacy Scale (S-GSE) is an instrument that measures perceived self-efficacy in problem-solving and goal achievement. The tool consists of 10 statements that are answered on a 4-point scale, ranging from 1 (not at all true) to 4 (exactly true). This scale is designed to assess an individual's belief in their ability to cope with a variety of difficult demands in life.
Depressive symtoms | Before surgery and 1, 3, and 6 months after surgery
  The Patient Health Questionnaire (PHQ-9) is a questionnaire that measures depressive symptoms. The form consists of 9 statements that are answered on a 4-point scale (0=not at all to 3=nearly every day). A total score of ≥ 10 indicates depressive symptoms.
Functional activity | Before surgery and 1, 3, and 6 months after surgery
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) is a tool that measures the level of functioning. The instrument consists of 12 questions that address difficulties related to health conditions, which are rated on a 5-point scale (1=no difficulty to 5=extreme difficulty/cannot do). A change of ≥5% compared to the baseline measurement indicates a clinically significant difference in the level of functioning.
Frailty | Before surgery and at 6 months after surgery
  The Clinical Frailty Scale (CFS) is an assessment scale of frailty consisting of nine levels (1=very fit to 9=terminally ill). The assessment is conducted by trained healthcare professionals by having the patient (or a relative) answer questions about their level of capacity two weeks prior.
Fatigue | Before surgery and at 6 months after surgery
  The Fatigue Scale for Motor and Cognitive Functions (FSMC) is a questionnaire that measures extreme forms of fatigue. The form consists of 20 statements concerning extreme fatigue and how it affects the participant's daily life and is answered on a 5-point scale (1= not true at all to 5= completely true). The FSMC measures both cognitive and physical fatigue. A total score of ≥ 43 indicates mild fatigue, ≥ 53 indicates moderate fatigue, and ≥ 63 indicates severe fatigue.
Health-related quality of life as assessed by RAND-36 | Before surgery and at 6 months after surgery
  RAND-36 is a questionnaire that measures health-related quality of life. The survey consists of 36 questions that assess 8 different domains of health: physical functioning, role limitations due to physical health, role limitations due to emotional problems, social functioning, emotional well-being, vitality, pain, and general health. Two different composite scores can be calculated for physical and mental health status, where a score of 50 or above indicates poor physical/mental health status.
Close relatives' assessment of cognition | Before surgery and 1, 3, and 6 months after surgery
  The Cognitive Failures Questionnaire for Others (f-CFQ) will be used to measure relatives' assessment of the patient's cognition. The instrument consists of 8 questions that assess the frequency of cognitive problems in daily life related to memory, attention, motor skills, and perception. The questions are answered on a 4-point scale ranging from (0=never to 4=very often).
Caregiver burden | Before surgery and 1, 3 and 6 months after surgery
  The Short Form Zarit Burden Interview (ZBI-12) will be used to measure caregiver burden. ZBI-12 consists of 12 questions that are answered on a 5-point scale (0=never to 4=almost always).
Experiences of cognitive recovery | At 6 months after surgery
  Qualitative semi-structured interviews
Close relatives experience | At 6 months after surgery
  Qualitative semi-structured interviews
Unplanned healthcare visits | At 6 months after surgery
  Study-specific questionnaire where participants will register any unplanned contacts or visits with healthcare services.

OTHER OUTCOMES:
Demographic and perioperative data | At baseline and perioperatively
  Will be collected from the medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Bergman L, Zecevic E, Damen T, Markovic G, Martinik A, Saarijarvi M, Eckerblad J, Nilsson U. Exploring cognitive function and postoperative neurocognitive recovery after cardiac surgery in older adults (ECPON): a protocol for an observational study. BMJ Open. 2025 Jun 22;15(6):e098208. doi: 10.1136/bmjopen-2024-098208. PMID 40545303